CLINICAL TRIAL: NCT02439099
Title: Retinoic Acid Homeostasis in Neuropsychiatric Diseases
Acronym: RAHND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Julian Hellmann-Regen, MD, Charite University, Berlin, Germany
Other Study IDs: EA4/002/13
Record Dates: First submitted 2015-04-02; First posted 2015-05-08 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Major Depression; Alzheimer's Disease; Alcoholism; Schizophrenia
MeSH Terms: conditions — Depressive Disorder, Major; Alzheimer Disease; Alcoholism; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral venous blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- MDD: Currently unmedicated patients with a depressive episode in the context of unipolar major depression
- Control: Healthy Controls
- Alzheimer's Disease: Patients with Alzheimer's disease
- Alcoholism: Subjects with alcoholism
- Schizophrenia: Subjects with before and schizophrenia prior to and during medication with clozapine, olanzapine or aripiprazole

SUMMARY:
It is hypothesized, that local retinoic acid (RA) homeostasis is functionally involved in the pathophysiology of depression. In a cross-sectional (and partly longitudinal) analysis, serum RA status will be assessed in healthy controls and subjects with Major Depression, Alzheimer's disease, alcoholism and in subjects with schizophrenia.

DETAILED DESCRIPTION:
Retinoids comprise of a group of small-molecule derivatives of Vitamin A with retinoic acid (RA) representing the biologically most active endogenous form. RA has multiple functions central nervous system (CNS). It is hypothesized, that local RA homeostasis is functionally involved in the pathophysiology of numerous neuropsychiatric diseases.

ELIGIBILITY:
MDD-Group

Inclusion Criteria:

* depressive episode in the context of unipolar major depression
* at least 18 points or more on the BDI and HAMD-17

Exclusion Criteria:

* additional or comorbid axis-I or axis-II disorder
* current history of any neurological or other serious medical condition
* any psychopharmacological treatment or substance use within the last two weeks or 5 half-lives (whichever is longer) of the respective substance
* any oral or topical application of retinoid-containing preparations within the last 3 months

AD-Group

Inclusion Criteria:

* diagnosed AD

Exclusion Criteria:

* any other neurodegenerative disorder
* any oral or topical application of retinoid-containing preparations within the last 3 months

Schizophrenia-Group

Inclusion Criteria:

* subjects with schizophrenia
* intended therapy with clozapine, olanzapine or aripiprazole
* BMI: 18 - 29,9 kg/m2

Exclusion Criteria:

* presence of diabetes or pathological glucose tolerance
* presence of and chronic inflammatory disease
* any psychopharmacological treatment of clozapine, olanzapine or aripiprazole within the last 3 months
* any oral or topical application of retinoid-containing preparations within the last 3 months

Alcoholism-Group

Inclusion Criteria:

* subjects with alcoholism who either still consume alcohol or are abstinent for at least 4 weeks

Exclusion Criteria:

* any oral or topical application of retinoid-containing preparations within the last 3 months
* current history of any neurological or other serious medical condition despite liver diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Out- and inpatients are eligible and will be recruited from patients seeking medical treatment at the Department of Psychiatry, Campus Benjamin Franklin, Charité, University Medicine Berlin.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Serum retinoic acid (RA) levels [nM] | Week 0
  Serum retinoic acid levels [nM] as determined by HPLC according to previously published protocols

SECONDARY OUTCOMES:
For MDD group: MADRS | Week 1, 3, 6
  Questionnaire to assess symptom severity in MDD
For MDD group: BDI II | Week 1, 3, 6
  Self-rating to assess of symptom severity in MDD
For MDD and schizophrenia Group: Change of serum retinoic acid (RA) levels [nM] | Week 1, 3, 6
  Serum retinoic acid levels [nM] as determined by HPLC according to previously published protocols
For schizophrenia group: Positive and Negative Syndrome Scale (PANSS) for Schizophrenia | Week 1, 3, 6
  Measurement of symptom severity of patients with schizophrenia
For schizophrenia group: Change of metabolic parametres For schizophrenia group:Positive and Negative Syndrome Scale (PANSS) | Week 1, 3, 6
  Assessmant of weight, blood pressure, levels of Glucose, HbA1c, cholesterols and dietry

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Heuser, MD, PhD, Principal Investigator — Chair: Department of Psychiatry, Charité, CBF
Locations (1):
- Department of Psychiatry, Charité - Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No